CLINICAL TRIAL: NCT01728077
Title: An Open-label, Multicenter, Follow-up Study to Evaluate the Long-term Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment in Subjects Aged 16 Years or Older With Epilepsy Phase 3b
Brief Title: Evaluation of Long-term Safety, and Efficacy of Brivaracetam (BRV) Used as Adjunctive Treatment in Subjects With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01372; 2012-000827-42 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2012-10-26; First posted 2012-11-16 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Long-term Follow-up; Epilepsy; Partial Onset Seizures; Adjunctive treatment
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): At Entry Visit (EV), subjects will start on the individualized Brivaracetam (BRV) dose that they had reached at the completion of the previous study. Dose adjustments of the Investigational Medicinal Product (IMP) are allowed at any time based on the clinical judgment of the investigator. The BRV dose can be increased or decreased in increments of 50 mg/day based on the individual subject's seizure control and/or tolerability; however, the BRV dose should not exceed 200 mg/day during the study and must always be administered as a symmetrical morning and evening dose. Upon completion or early discontinuation from this study, there will be a Down-Titration Period in steps of 50 mg/day on a weekly basis until 20 mg/day for 1 week is reached, followed by a Post-Treatment Period (between 2 and 4 weeks) during which the subject will not receive study drug. No down-Titration Period will be applicable if subjects are continued on BRV after they complete this study.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Flexible dosing, can up and down-titrate as needed.
  Other Names: UCB34714

SUMMARY:
N01372 study is to evaluate the long-term safety, tolerability, maintenance of efficacy of Brivaracetam (BRV); as well as the effect of BRV on subjects' health-related quality of life and to explore the direct medical resource use for BRV (for subjects entering N01372 from a study where pharmacoeconomic data was collected). BRV will be used at doses up to maximum of 200 mg/day, as adjunctive treatment in subjects aged 16 years or older with Epilepsy.

DETAILED DESCRIPTION:
Flexible dosing up to 200 mg/day, twice daily (10, 25 and 50 mg oral film-coated tablets). The study will continue until either regulatory approval of BRV has been granted by any Health Authority in an indication of adjunctive treatment of Epilepsy, or until the Sponsor decides to close the study, or until the BRV development is stopped by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and 16 years or older. Subjects under 18 years of age may be included only where legally permitted and ethically accepted
* Subjects having completed the Treatment Period of an applicable previous BRV study, and have access to the present study
* Subject for whom the investigator believes a reasonable benefit from the long-term administration of BRV may be expected
* Female subjects without childbearing potential (postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible. Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method
* Subjects must be able to take the oral film-coated tablets of BRV

Exclusion Criteria:

* Subject has developed hypersensitivity to any components of the Investigational Medicinal Product (IMP) or comparative drugs as stated in the protocol during the course of the prior study
* Severe medical, neurological, or psychiatric disorders, or laboratory values that may have an impact on the safety of the subject
* Poor compliance with the visit schedule or medication intake in the previous BRV study
* Planned participation in any other clinical study of another investigational drug or device during this study
* Pregnant or lactating woman
* Any medical condition which, in the investigator's opinion, warrants exclusion
* Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either question 4 or question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at the last visit of the previous study or at the Entry Visit of this study if not completed at the last visit of the previous study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (10):
- United States (6):
  - 103, Little Rock, Arkansas
  - 108, Lexington, Kentucky
  - 109, New York, New York
  - 106, Akron, Ohio
  - 110, Dallas, Texas
  - 102, Salt Lake City, Utah
- 201, Paris, France
- Germany (2):
  - 303, Bernau
  - 300, Kehl-Kork
- 502, Seville, Spain

REFERENCES:
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in October 2012 and concluded in August 2016.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS), which consisted of all subjects who took at least 1 dose of study drug.
Groups:
- Brivaracetam Focal Epilepsy: This arm includes subjects with focal epilepsy, who received a flexible dose of Brivaracetam (BRV) tablets, administered twice a day, starting with an individual dose that they had reached at the completion of study N01395 (feeder study). The BRV dose could have been increased or decreased in increments of 50mg/day based on the individual subject's seizure control and/or tolerability, but was to not exceed 200mg/day.
- Brivaracetam Generalized Epilepsy: This arm includes subjects with generalized epilepsy, who received a flexible dose of Brivaracetam (BRV) tablets, administered twice a day, starting with an individual dose that they had reached at the completion of study N01395 (feeder study). The BRV dose could have been increased or decreased in increments of 50mg/day based on the individual subject's seizure control and/or tolerability, but was to not exceed 200mg/day.
Period: Overall Study
Arm/Group | Brivaracetam Focal Epilepsy | Brivaracetam Generalized Epilepsy
Started | 19 | 7
Completed | 11 | 2
Not Completed | 8 | 5
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject choice | 2 | 3
Not completed — Death | 0 | 1
Not completed — Patient moving | 1 | 0
Not completed — Non compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set, which consisted of all subjects who received at least 1 dose of study medication.
Arm/Group | Brivaracetam Focal Epilepsy | Brivaracetam Generalized Epilepsy | Total Title
Number analyzed (Participants) | 19 | 7 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 7 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Arithmetic mean (standard deviation) | 38.6 (10.9) | 30.7 (13.2) | 36.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 12 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs) During Evaluation Period
Description: TEAEs were defined as AEs that had onset on or after the day of first study medication dose. An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. Results are presented as the percentage of subjects with at least one treatment-emergent adverse event during this study.
Time Frame: From Entry Visit (Month 0) to the Last Evaluation Period Visit or Early Discontinuation Visit (up to 46 months)
Measure: Number; unit: percentage of subjects
Groups:
- Brivaracetam Focal Epilepsy (SS): This arm includes subjects with focal epilepsy, who received a flexible dose of Brivaracetam (BRV) tablets, administered twice a day, starting with an individual dose that they had reached at the completion of study N01395 (feeder study). The BRV dose could have been increased or decreased in increments of 50mg/day based on the individual subject's seizure control and/or tolerability, but was to not exceed 200mg/day. This arm is part of the Safety Set (SS).
- Brivaracetam Generalized Epilepsy (SS): This arm includes subjects with generalized epilepsy, who received a flexible dose of Brivaracetam (BRV) tablets, administered twice a day, starting with an individual dose that they had reached at the completion of study N01395 (feeder study). The BRV dose could have been increased or decreased in increments of 50mg/day based on the individual subject's seizure control and/or tolerability, but was to not exceed 200mg/day. This arm is part of the Safety Set (SS).
Arm/Group | Brivaracetam Focal Epilepsy (SS) | Brivaracetam Generalized Epilepsy (SS)
Number analyzed (Participants) | 19 | 7
percentage of subjects | 78.9 | 71.4

2. Primary Outcome: Percentage of Subjects Withdrawn Due to an Adverse Event (AE) During the Evaluation Period
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. Results are presented as the percentage of subjects withdrawn due to an AE.
Time Frame: From Entry Visit (Month 0) to the Last Evaluation Period Visit or Early Discontinuation Visit (up to 46 months)
Measure: Number; unit: percentage of subjects
Arm/Group | Brivaracetam Focal Epilepsy (SS) | Brivaracetam Generalized Epilepsy (SS)
Number analyzed (Participants) | 19 | 7
percentage of subjects | 0 | 14.3

3. Primary Outcome: Occurrence of a Serious Adverse Event (SAE) During the Evaluation Period
Description: SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity or are a congenital anomaly/birth defects. Results are presented as the percentage of subjects with at least one SAE during this study.
Time Frame: From Entry Visit (Month 0) to the Last Evaluation Period Visit or Early Discontinuation Visit (up to 46 months)
Population: The analysis was performed on the Safety Set (SS), which consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | Brivaracetam Focal Epilepsy (SS) | Brivaracetam Generalized Epilepsy (SS)
Number analyzed (Participants) | 19 | 7
percentage of subjects | 26.3 | 28.6

4. Secondary Outcome: Frequency of Partial-Onset Seizure (POS) Type I Per 28 Days During the Evaluation Period for Subjects With Focal-onset Epilepsy
Description: The POS frequency is standardized to a 28-day duration. Results are presented as the median number of seizures per 28 days.
Time Frame: From Entry Visit (Month 0) to the Last Evaluation Period Visit or Early Discontinuation Visit (up to 46 months)
Population: The analysis was performed on the Efficacy Analysis Set (EAS), which consisted of subjects who took at least one dose of study drug and had at least one seizure daily record card (DRC) day during the Evaluation Period.
Measure: Median (Full Range); unit: Seizures per 28 days
Groups:
- Brivaracetam Focal Epilepsy (EAS): This arm includes subjects with focal epilepsy, who received a flexible dose of Brivaracetam (BRV) tablets, administered twice a day, starting with an individual dose that they had reached at the completion of study N01395 (feeder study). The BRV dose could have been increased or decreased in increments of 50mg/day based on the individual subject's seizure control and/or tolerability, but was to not exceed 200mg/day. This arm is part of the Efficacy Analysis Set (EAS).
Arm/Group | Brivaracetam Focal Epilepsy (EAS)
Number analyzed (Participants) | 17
Seizures per 28 days | 0.4 [0 to 124]

5. Secondary Outcome: Percentage of Change in Partial-Onset-Seizure (POS) Type I Frequency Per 28 Days From Baseline of the Previous Study to the Evaluation Period for Subjects With Focal-onset Epilepsy Entering N01372 From a Study Where Baseline Seizure Data Was Collected
Description: The POS frequency is standardized to a 28-day duration. Results are presented as the median percentage of reduction per 28 days. Negative values indicate improvement from Baseline.
Time Frame: From Baseline of the previous study to the Last Evaluation Period Visit or Early Discontinuation Visit (up to 49 months)
Population: as for outcome 4
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Brivaracetam Focal Epilepsy (EAS)
Number analyzed (Participants) | 17
percentage of change | -56.3 [-97 to 717]

6. Secondary Outcome: 50 % Responder Rate in Partial-Onset-Seizure (POS) Type I Frequency From Baseline of the Previous Study to the Evaluation Period for Subjects With Focal-onset Epilepsy Entering N01372 From a Study Where Baseline Seizure Data Was Collected
Description: The POS frequency is standardized to a 28-day duration. A responder is defined as a subject with a >=50% reduction in seizure frequency from the Baseline Period of the previous study. Results are presented as the percentage of subjects with 50 % responder rate in POS Type I frequency.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Brivaracetam Focal Epilepsy (EAS)
Number analyzed (Participants) | 17
percentage of subjects | 54.5

ADVERSE EVENTS:
Time Frame: Adverse events collection started at Day 0 and continued up to 30 days after last intake of study medication.
Arm/Group | Brivaracetam Focal Epilepsy (SS) | Brivaracetam Generalized Epilepsy (SS)
Serious Adverse Events (participants affected / at risk) | 5/19 | 2/7
Other Adverse Events (participants affected / at risk) | 13/19 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam Focal Epilepsy (SS) (N=19) | Brivaracetam Generalized Epilepsy (SS) (N=7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (3) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam Focal Epilepsy (SS) (N=19) | Brivaracetam Generalized Epilepsy (SS) (N=7)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (3)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract (Infections and infestations) | 1 (1) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (4) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Crystal urine present (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 2 (3) | 0 (0)
Protein urine present (Investigations) | 2 (3) | 0 (0)
Urinary casts (Investigations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Headache (Nervous system disorders) | 7 (68) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (29) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (20) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days